CLINICAL TRIAL: NCT07336771
Title: A Multicenter, Open-Label, Phase Ib/II Randomized Study of JSKN016 in Combination With D-0502 in Patients With Locally Advanced or Metastatic Hormone Receptor-Positive, HER2-Negative Breast Cancer
Brief Title: JSKN016 in Combination With D-0502 for Locally Advanced or Metastatic HR-Positive, HER2-Negative Breast Cancer
Status: Not yet recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Jiangsu Alphamab Biopharmaceuticals Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: JSKN016-204
Record Dates: First submitted 2025-12-23; First posted 2026-01-13 (Actual); Last update posted 2026-01-13 (Actual); Status verified 2026-01

CONDITIONS: Metastatic Breast Cancer; Locally Advanced Breast Cancer (LABC)
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- JSKN016 Q2W + D-0502 (Experimental)
  Interventions: Drug: JSKN016 Q2W; Drug: D-0502
- JSKN016 Q3W + D-0502 (Experimental)
  Interventions: Drug: JSKN016 Q3W; Drug: D-0502

INTERVENTIONS:
Drug: JSKN016 Q2W — 4 mg/kg, intravenous infusion, every 2 weeks
  Arms: JSKN016 Q2W + D-0502
Drug: JSKN016 Q3W — 4 mg/kg, intravenous infusion, every 3 weeks
  Arms: JSKN016 Q3W + D-0502
Drug: D-0502 — 200 mg, oral, once daily

SUMMARY:
This is a multicenter, open-label, Phase Ib/II randomized study designed to evaluate the safety, tolerability, dose-limiting toxicities (DLTs), and preliminary antitumor activity of JSKN016 in combination with the oral selective estrogen receptor degrader (SERD) D-0502 in patients with locally advanced or metastatic hormone receptor-positive (HR+), HER2-negative breast cancer who have previously progressed on CDK4/6 inhibitor-based endocrine therapy.

Approximately 60 patients will be randomized in a 1:1 ratio to receive JSKN016 administered intravenously every 2 weeks (Q2W) or every 3 weeks (Q3W), in combination with daily oral D-0502. Each dosing cohort will include a safety lead-in phase to assess DLTs prior to cohort expansion. Tumor response will be assessed according to RECIST v1.1.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years
* Histologically or cytologically confirmed locally advanced or metastatic HR-positive, HER2-negative breast cancer
* HR-positive defined as ER and/or PR ≥1% by IHC
* HER2-negative per ASCO/CAP guidelines
* At least one measurable extracranial lesion per RECIST v1.1
* ECOG performance status 0-1
* Prior progression on CDK4/6 inhibitor plus endocrine therapy
* Adequate organ and cardiac function
* Postmenopausal women, or premenopausal women receiving ovarian function suppression

Exclusion Criteria:

* Active or untreated CNS metastases
* Prior treatment with ADCs containing topoisomerase I inhibitor payloads
* Active interstitial lung disease or pneumonitis
* Uncontrolled cardiovascular disease or active infection
* Prior malignancy within 5 years (with specific exceptions)
* Pregnancy or breastfeeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2027-12 (Estimated); Study Completion 2028-06 (Estimated)

PRIMARY OUTCOMES:
Incidence of dose-limiting toxicities (DLTs) | From first dose through the end of Cycle 1 (approximately 21 days)
Objective Response Rate (ORR) | From first dose through treatment discontinuation, assessed up to 12 months
Safety and tolerability (TEAEs, TRAEs, SAEs) | From first dose until 30 days after the last dose of study treatment.

SECONDARY OUTCOMES:
Disease Control Rate (DCR) | From first dose through 24 weeks
Duration of Response (DoR) | From first documented objective response (CR or PR) until disease progression or death, whichever occurs first, assessed up to 24 months
Clinical Benefit Rate (CBR) | From first dose through 24 weeks
Progression-Free Survival (PFS) | From first dose until the first documented disease progression or death from any cause, whichever occurs first, assessed up to 24 months
Overall Survival (OS) | From first dose until death from any cause, assessed up to 36 months

CONTACTS AND LOCATIONS:
Locations (1):
- Fudan University Shanghai Cancer center, Shanghai, China

IPD SHARING:
Plan to Share IPD: No